CLINICAL TRIAL: NCT03713021
Title: Evaluation of TraceIT Tissue Marker to Mark the Primary Resection Bed Margins of Oropharyngeal Cancers: a Pilot Study
Brief Title: TraceIT Tissue Marker to Mark the Primary Resection Bed Margins of Oropharyngeal Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment unavailable
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201810117
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TraceIT Tissue Marker (Experimental): * Following successful tumor resection, TraceIT Tissue Marker will be applied in 0.2 to 0.5 mL injections at 5 locations to mark the tumor bed: superiorly, inferiorly, laterally, medially, and center of resection. The marginal injections will be within 3 mm of the resection edge and within 5 mm deep. The center of the resection bed will be injected within 5 mm deep if possible.
  * Within 6 weeks after surgery, a CT simulation scan will be performed per normal protocol for patients receiving surgery followed by adjuvant therapy. This scan will be used to generate the intensity-modulated radiation therapy (IMRT) treatment plan
  * Two treatment plans will be performed per patient using the simulation CT scan. One will be the standard of care treatment plan and will be the basis of the actual radiation treatment they receive. The second treatment plan will be based on utilizing the TraceIT hydrogel markers as a guide for the resection bed.
  Interventions: Device: TraceIT Tissue Marker

INTERVENTIONS:
Device: TraceIT Tissue Marker — The maximum injection volume of TraceIT hydrogel, for a single location, is 1mL.
  Other Names: TraceIT hydrogel

SUMMARY:
The purpose of this research study is to look at how using an injectable marker called TraceIT can help with the radiation treatment planning process. TraceIT is a gel that dissolves in the body over time and can be injected and is visible on many types of images that can be used in the treatment planning process. If the exact edges of negative tumor margins can be marked before treatment planning, it is thought that the area receiving radiation can be more personalized, thus potentially reducing unnecessary radiation to areas that are cancer-free.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed (by routine H&E staining) or highly suspicious for oropharyngeal squamous cell cancer.
* Planned treatment includes transoral surgery followed by adjuvant intensity modulated radiation therapy (IMRT).
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Distant metastatic disease at the time of definitive treatment, and thus study, initiation.
* History of major head & neck surgery or previous head & neck irradiation.
* History of or current oral disease that may interfere with interpretation of study outcomes.
* Currently enrolled in another radiation therapy trial that has not completed its primary endpoint or that clinically interferes with this study.
* Poor surgical candidate
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan S Jackson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TraceIT Tissue Marker
Started | 27
Completed | 12
Not Completed | 15
Not completed — Did not have CT sim scan available | 6
Not completed — Not eligible | 4
Not completed — Issues with TraceIT markers | 5

BASELINE CHARACTERISTICS:
Arm/Group | TraceIT Tissue Marker
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Mean Clinical Target Volumes (CTV) Between the Standard of Care Treatment Plan and the Treatment Plan Based on the TraceIT Hydrogel Markers
Description: -The mean total dose of each targeted site was totaled from the standard of care treatment plan and the TraceIT tissue marker treatment plan. The percent change in CTV was measured by standard field in cGy minus marker based in cGy = percent change in CTV (in cGy). The sites included left & right submandibular, left & right parotid, left & right pharynx constrictor, oral cavity, lips, larynx, and spinal cord.
Time Frame: At the treatment planning (2-5 weeks after TraceIT hydrogel placement)
Population: 12 participants had both standard of care treatment plans and TraceIT tissue marker treatment plans available for this outcome measure.
Measure: Number; unit: percent change in total CTV
Arm/Group | TraceIT Tissue Marker
Number analyzed (Participants) | 12
percent change in total CTV
  Subject 001: number analyzed (Participants) | 1
  Subject 001 | 54.35
  Subject 002: number analyzed (Participants) | 1
  Subject 002 | 54.07
  Subject 003: number analyzed (Participants) | 1
  Subject 003 | -30.40
  Subject 004: number analyzed (Participants) | 1
  Subject 004 | 50.95
  Subject 005: number analyzed (Participants) | 1
  Subject 005 | 53.63
  Subject 006: number analyzed (Participants) | 1
  Subject 006 | 62.53
  Subject 007: number analyzed (Participants) | 1
  Subject 007 | 54.30
  Subject 008: number analyzed (Participants) | 1
  Subject 008 | 60.65
  Subject 009: number analyzed (Participants) | 1
  Subject 009 | 32.96
  Subject 010: number analyzed (Participants) | 1
  Subject 010 | 45.51
  Subject 011: number analyzed (Participants) | 1
  Subject 011 | 29.50
  Subject 012: number analyzed (Participants) | 1
  Subject 012 | 17.60

2. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event Related to TraceIT Injection
Time Frame: From time of injection through surgery (day 1)
Population: 14 out of the enrolled 27 participants received the TraceIT marker and were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TraceIT Tissue Marker
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Anatomic Localization Related to Standard Treatment Fields Based on Anatomy as Measured by Number of Participants That Had Markers Visible
Time Frame: At the treatment planning (2-5 weeks after TraceIT hydrogel placement)
Population: 21 out of 27 participants had CT sim scans available.
Measure: Count of Participants; unit: Participants
Arm/Group | TraceIT Tissue Marker
Number analyzed (Participants) | 21
Participants | 15

ADVERSE EVENTS:
Time Frame: Adverse events were followed from time of TraceIT injection through the intraoperative period (day 1).
Description: 14 out of 27 participants enrolled received the TraceIT marker. All-cause mortality, serious adverse event and adverse event data were collected on those patients who received the TraceIT marker.
Arm/Group | TraceIT Tissue Marker
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03713021/Prot_SAP_000.pdf